CLINICAL TRIAL: NCT02337972
Title: Conjunctival Flora Patterns After Serial Intravitreal Injections Without Postinjection Topical Antibiotics in Diabetic Patients
Brief Title: Conjunctival Flora Patterns After Serial Intravitreal Injections in Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Irina Barequet, Head of cornea unit, Ophthalmology department, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Sheba_Medical_Center
Record Dates: First submitted 2015-01-01; First posted 2015-01-14 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Diabetic Retinopathy; Diabetic Macular Edema
Keywords: diabetic macular edema; Intravitreal injection; conjunctival flora
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diabetic patients (Experimental): Patients with Diabetes Mellitus and macular edema who were determined by their treating physician to require at least 3 serial injections with an anti-Vascular epithelial growth factor (VEGF). Prior to each injection a use of povidone-iodine 4% drops will be performed to clean the conjunctival sac
  Interventions: Drug: povidone-iodine 4%

INTERVENTIONS:
Drug: povidone-iodine 4% — Prior to each injection and before the use of povidone-iodine drops, a conjunctival culture will be taken
  Other Names: Wokadine; Pyodine

SUMMARY:
The aim of this study is to investigate the conjunctival bacterial flora and antibiotic resistance patterns following serial intravitreal injections of anti-VEGF in diabetic patients, using a povidone-iodine preparation without preinjection or postinjection topical antibiotics.

DETAILED DESCRIPTION:
The study is designed to enroll patients with Diabetes Mellitus over 18 years of age with diagnosis of diabetic retinopathy and diabetic macular edema, who were determined by their treating physician to require at least 3 serial injections with an anti-VEGF agent.

After signing an informed consent, conjunctival cultures will be performed from the participants' both eyes at baseline and at each subsequent injection. Prior to each injection and the use of povidone-iodine drops, a conjunctival culture will be taken by swabbing the inferior fornix. Another culture will be taken twenty minutes after the injection. We will culture the swab samples on blood and chocolate agar plates.

All patients will be asked to complete a questionnaire regarding their signs and symptoms after the injection (like burning sensation, itching, discharge, tearing etc). The following routine procedure will be used in all intravitreal injections: local anesthesia using Oxybuprocaine hydrochloride, ocular surface and eyelids sterilization with topical povidone-iodine 4%. Intravitreal injection of 3.5 mm will be performed posterior to the limbus in pseudophakic patients and 4 mm injection will be performed posterior to the limbus in phakic patients using a 30 gauge needle.

The exclusion criteria will consist patients who had received a prior intraocular injection in either eye, current use of contact lenses, chronic use of any ophthalmic medication, ocular surgery within the past 6 months, use of systemic antibiotics within the past 6 months and known allergy or contraindication to povidone-iodine or proparacaine.

The study is planned to enroll 50 patients.

ELIGIBILITY:
Inclusion Criteria:

* age above 18
* patients with diabetes mellitus
* patients with diabetic macular edema

Exclusion Criteria:

* patients who had received a prior intraocular injection in either eye,
* current use of contact lenses,
* chronic use of any ophthalmic medication,
* ocular surgery within the past 6 months,
* use of systemic antibiotics within the past 6 months,
* known allergy or contraindication to povidone-iodine or proparacaine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Change of conjunctival flora and bacterial resistance | 4 month

CONTACTS AND LOCATIONS:
Overall Officials: Irit Barequet, MD, Principal Investigator — Sheba medical center, Ophthalmology department
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Non-US Resident, Israel